CLINICAL TRIAL: NCT05492656
Title: Accuracy and Feasibility of CADx System for White Light Colonic Polyp Characterization
Brief Title: Accuracy of CADx System for White Light Colonic Polyp Characterization
Acronym: GIC
Status: Completed | Type: Observational
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Franco Radaelli, Head of Gastroenterology Unit, Valduce Hospital
Other Study IDs: 41/2022
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Colonic Polyp; Adenoma Colon
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The endoscopist performances in the optical diagnosis (OD) of colonic polyps with the available technologies vary widely across centers and across endoscopists. The OD process is strictly related to the operator training and expertise. Most of the available studies in optical characterization have been carried out by expert endoscopist in tertiary high volume centers, and weren't replied on large unselected populations. For these reasons, at the moment the optical characterization of polypoid lesions can't replace, in the everyday clinical practice, the histopathological evaluation of resected polyps. Artificial intelligence (AI)-based systems have the potential to make optical characterization process of colonic polyps easier and more reliable, thus supporting the endoscopist in the application of leave-in-situ and of resect-and-discard strategies. The implementation of such strategies would lead to a significant economic saving and a decrease of risks and complications related to unnecessary polypectomy. GI-Genius System (Medtronic Inc, Minneaopolis, USA) is a CNN-based algorithm allowing an automatic OD of colonic polyps. This system does not require dedicated light setting for polyp evaluation as it works with white light high definition images, which are the actual standard in every endoscopic unit. During colonoscopy, when a polyp is framed within the screen, a green detection box surrounds the polyp and the system automatically provides (whenever possible) the optical diagnosis labeling the polyp as "adenoma or non-adenoma". When the automatic polyp charaterization is unfeasible the label "no prediction" appears. Nowadays only few data about the feasibility and performances of this system in clinical practice are available. In addition published studies are mostly focused on technical rather thann clinical issues. The present prospective observational trial is primarily aimed at evaluating the diagnostic accuracy of optical characterization of colonic polyps <= 1 cm using GI-Genius System in daily clinical practice, having histopathology examination as reference standard.

ELIGIBILITY:
Inclusion Criteria:

Consecutive outpatients undergoing colonoscopy for one of the following indication:

* FIT-based screening program
* voluntary screening
* post-polipectomy surveillance
* gastrointestinal symptoms
* family history of colorectal cancer.

Exclusion Criteria:

* urgent colonoscopy
* patients in which polyps could not be resected (e.g ongoing anticoagulation therapy)
* patients with past colorectal cancer or polyposis syndrome

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adults (18-85 years) outpatients referred for colonoscopy are invited to participate in the present study.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CADx in evaluating small colonic polyps | Entire study duration (3 months)
  Numer of correctly characterized polyps using AI/total number of detected polyps

SECONDARY OUTCOMES:
Feasibility of CADx in evaluating small colonic polyps | Entire study duration (3 months)
  Number of characterizable polyps using AI/total number of detected polyps
Sensitivity | Entire study duration (3 months)
  CADx sensitivity (rate of TP/TP+FN) will be calculated having histopathology as reference standard and according to polyp size and location
specificity | Entire study duration (3 months)
  CADx specificity (rate of TN/TN+FP) will be calculated having histopathology as reference standard according to polyp size and location
Positive predictive value | Entire study duration (3 months)
  CADx positive predictive value (rate of TP/TP+FP) will be calculated having histopathology as reference standard according to polyp size and location
Negative predictive value | Entire study duration (3 months)
  CADX negative predictive value (rate of TN/TN+FN) will be calculated having histopathology as reference standard according to polyp size and location

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Unit, Valduce Hospital, Como, Italy

IPD SHARING:
Plan to Share IPD: Undecided